CLINICAL TRIAL: NCT00629746
Title: Intraoperative Electromyographic Monitoring of the Recurrent Laryngeal Nerve in Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Feng-Yu Chiang, MD, Department of Otolaryngology, Kaohsiung Medical University, Taiwan.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMUH-IRB-EMG-01
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-05

CONDITIONS: Thyroid Surgery; Recurrent Laryngeal Nerve; Electromyographic Monitoring
Keywords: Thyroid; RLN; EMG
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NIM (Nerve Integrity Monitor) (Experimental)
  Interventions: Device: Medtronic Xomed Nerve Integrity Monitor (NIM)

INTERVENTIONS:
Device: Medtronic Xomed Nerve Integrity Monitor (NIM) — patients receive surgery will be intubated with Medtronic Xomed NIM EMG endotracheal tube and the device will be connected to the monitoring system
  1. The channel leads from the NIM EMG reinforced endotracheal tube were connected to a NIM-response monitor
  2. A Prass monopolar probe was used in direct contact with the vagus nerve and RLN for laryngeal nerve stimulation.
  3. The stimuli were generated from the NIM-Response monitor for vagal and RLN stimulation.
  4. The NIM-response monitor was set to run with a 50 millisecond time window and an amplitude scale at 0.2 mV/division. Event capture was activated with a threshold at 100 μV. Peak to peak amplitudes of evoked EMG activities were directly read on the monitor screen.
  Other Names: (Medtronic Xomed, Jacksonville, FL).

SUMMARY:
The purpose of this study will explore the advantages of electrodes used for monitoring of the recurrent laryngeal nerve (RLN) in thyroid surgery

DETAILED DESCRIPTION:
OBJECTIVES/HYPOTHESIS:

The purpose of this study will explore the advantages and applications of electrodes used for monitoring of the recurrent laryngeal nerve (RLN) in thyroid surgery. We want to know that if the monitoring system will decrease the rate of recurrent laryngeal nerve palsy.

STUDY DESIGN:

One hundred patients who undergoing thyroid surgery will be collected in this study. Patients will be intubated for general anesthesia with a Medtronic Xomed Nerve Integrity Monitor (NIM) EMG endotracheal tube (Jacksonville, Fla) that had 2 electrodes imbedded in the wall of the endotracheal tube. These wires were placed up against each vocal cord. Two grounding wires(needle No. 26) were placed up in the subcutaneous tissues of both shoulders. The electrode wires, grounding wires, and nerve stimulator were connected to a monitoring device (Medtronic NIM-Response) that recoded a visual evoked potential and audible beep to each muscle contraction of a vocal cord. A Medtronic Xomed Prass monopolar nerve stimulator wand was used to test the RLN intraoperatively and was set at 0.5mA. Direct physical touching of the RLN with nerve stimulator using pulsed current would produce an audible "beep-beep-beep".

CONCLUSION:

This study will be conducted in cooperation with Department of anesthesiology. The following subjects will be collected and elucidated:

1. If the muscle relaxant used during surgery will affect the operation of RLN monitoring system.
2. Can RLN monitoring system accurately identify the RLN
3. Can RLN monitoring system accurately predict the function of RLN
4. Can RLN monitoring system decrease the RLN palsy rate after thyroidectomy
5. Application of RLN monitoring to determine the safety and the benefit of vagal stimulation at the beginning and the end of thyroid operation
6. Application of RLN monitoring to determine whether extensive dissection of RLN increases the risk of nerve injury.

At least four papers will be written after this study with the topics as followings:

1. Influence of muscle relaxation on neuromonitoring of the recurrent laryngeal nerve during thyroid surgery
2. Intraoperative neuromonitoring of the recurrent laryngeal nerve during thyroid surgery: Plaudits and pitfalls 3. Vagal stimulation during intraoperative neuromonitoring of the recurrent laryngeal nerve in thyroid operation.

4. Does extensive dissection of recurrent laryngeal nerve during thyroid operation increase the risk of nerve injury? Our experience with the application of intraoperative neuromonitoring

ELIGIBILITY:
Inclusion Criteria:

* Thyroid disease for operation

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
If the muscle relaxant used during surgery will affect the operation of RLN monitoring system. | during operation

SECONDARY OUTCOMES:
Can RLN monitoring system accurately predict the function of RLN Can RLN monitoring system decrease the RLN palsy rate after thyroidectomy | early postoperation period
Can standardization of IONM procedures further lower the RLN palsy rate | early postoperation period
Dose IONM help to decrease the RLN palsy rate during difficult thyroid operations | early postoperation period

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Yu Chiang, M.D., Study Director — Department of Otolaryngology- Head and Neck Surgery, Kaohsiung Medical University Hospital, Kaohsiung Medical University, Taiwan; Che-Wei Wu, MD, Principal Investigator — Department of Otolaryngology- Head and Neck Surgery,Kaohsiung Medical University Hospital, Kaohsiung Medical University, Taiwan
Locations (1):
- Department of Otolaryngology- Head and Neck Surgery, Kaohsiung Medical University Hospital, Kaohsiung Medical University, Taiwan, Kaohsiung City, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Wu CW, Dionigi G, Chen HC, Chen HY, Lee KW, Lu IC, Chang PY, Hsiao PJ, Ho KY, Chiang FY. Vagal nerve stimulation without dissecting the carotid sheath during intraoperative neuromonitoring of the recurrent laryngeal nerve in thyroid surgery. Head Neck. 2013 Oct;35(10):1443-7. doi: 10.1002/hed.23154. Epub 2012 Sep 18. PMID 22987562
- [Derived] Chiang FY, Lu IC, Tsai CJ, Hsiao PJ, Lee KW, Wu CW. Detecting and identifying nonrecurrent laryngeal nerve with the application of intraoperative neuromonitoring during thyroid and parathyroid operation. Am J Otolaryngol. 2012 Jan-Feb;33(1):1-5. doi: 10.1016/j.amjoto.2010.11.011. Epub 2011 Feb 8. PMID 21306793
- [Derived] Chiang FY, Lu IC, Tsai CJ, Hsiao PJ, Hsu CC, Wu CW. Does extensive dissection of recurrent laryngeal nerve during thyroid operation increase the risk of nerve injury? Evidence from the application of intraoperative neuromonitoring. Am J Otolaryngol. 2011 Nov-Dec;32(6):499-503. doi: 10.1016/j.amjoto.2010.11.001. Epub 2011 Feb 8. PMID 21306792
- [Derived] Chiang FY, Lu IC, Chen HC, Chen HY, Tsai CJ, Lee KW, Hsiao PJ, Wu CW. Intraoperative neuromonitoring for early localization and identification of recurrent laryngeal nerve during thyroid surgery. Kaohsiung J Med Sci. 2010 Dec;26(12):633-9. doi: 10.1016/S1607-551X(10)70097-8. PMID 21186011
- [Derived] Chiang FY, Lu IC, Kuo WR, Lee KW, Chang NC, Wu CW. The mechanism of recurrent laryngeal nerve injury during thyroid surgery--the application of intraoperative neuromonitoring. Surgery. 2008 Jun;143(6):743-9. doi: 10.1016/j.surg.2008.02.006. PMID 18549890